CLINICAL TRIAL: NCT01500772
Title: A Multicenter, Single-arm Trial Evaluating the Safety and Efficacy of DEB025/Alisporivir in Combination With Pegylated Interferon-α2a and Ribavirin (Peg-IFNα2a/RBV) in Protease Inhibitor Treatment Failure Patients With Chronic Hepatitis C Genotype 1
Brief Title: Alisporivir With PEG and RBV in Protease Inhibitor (PI) Treatment Failure Patients With Chronic Hepatitis C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2306; 2011-004653-31 (EudraCT Number)
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; PI treatment failure
MeSH Terms: conditions — Hepatitis C | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

ARMS (1):
- Alisporivir (Experimental): ALV 400 mg twice daily (BID), plus PEG and RBV for 48 weeks
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Alisporivir — ALV 200 mg soft gel capsules administered orally
  Other Names: DEB025
Drug: Peginterferon alfa-2a — PEG 180 μg administered via subcutaneous (s.c.) injection once weekly
  Other Names: Pegasys®
Drug: Ribavirin — RBV 200 mg tablets (weight-based dose: < 75 mg = 1000 mg/day; ≥ 75 kg = 1200 mg/day) administered orally in a divided daily dose
  Other Names: Copegus®; RBV

SUMMARY:
This study is to evaluate the overall efficacy, and safety profile of the triple combination therapy of alisporivir (ALV; DEB025) plus peginterferon alfa-2a (PEG) and ribavirin (RBV) patients with chronic hepatitis C (HCV) genotype 1 who failed prior treatment with a protease inhibitor (PI).

ELIGIBILITY:
Inclusion criteria:

1. Patients with chronic HCV genotype 1 infection with previous PI treatment failure
2. Three months minimum time from the last dose of previous PI treatment to the first dose of study medication

Exclusion criteria:

1. Use of other investigational drugs at the time of enrollment
2. History of hypersensitivity to PEG or RBV
3. Any null non-responders to prior PEG/RBV treatment

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (23):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigational site, Bradenton, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Brockton, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Alexandria, Virginia
  - Novartis Investigative Site, Newport News, Virginia
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- France (3):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Germany (14):
  - Novartis Investigational Site, Berlin
  - Novartis Investigative Site, Berlin
  - Novartis Investigational Site, Cologne
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigational Site, Frieburg
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigational Site, Mainz
  - Novartis Investigative Site, Mainz
- Italy (8):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bologna
- Novartis Investigative Site, San Juan, Puerto Rico
- Spain (2):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Majadanonda, Madrid
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Alisporivir: Alisporivir (ALV) 400 mg twice daily (BID), with peginterferon alfa-2a (PEG) and ribavirin (RBV) for 48 weeks.
Period: Overall Study
Arm/Group | Alisporivir
Started | 6
Completed | 0
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Alisporivir: ALV 400 mg BID with PEG and RBV for 48 weeks.
Arm/Group | Alisporivir
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sustained Viral Response (SVR) 12 Weeks After End of Treatment (SVR12)
Description: SVR12 was defined as hepatitis C (HCV) ribonucleic acid (RNA) laboratory value below level of quantification (LOQ) (i.e., 25 IU/ml) 12 weeks after the end of treatment.
Time Frame: 12 weeks posttreatment
Population: The study was terminated before the outcome measure time point.
Arm/Group | Alisporivir
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants Who Achieved SVR 24 Weeks After the End of Treatment (SVR24)
Description: SVR24 was defined as HCV RNA laboratory value < LOQ 24 weeks after the end of treatment.
Time Frame: 24 weeks posttreatment
Population: The study was terminated before the outcome measure time point.
Arm/Group | Alisporivir
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA Laboratory Value Below Level of Detection 12 Weeks After the End of Treatment (SVR12-LOD)
Description: Level of detection (LOD) was defined as 10 IU/mL
Time Frame: 12 weeks posttreatment
Population: The study was terminated before the outcome measure time point.
Arm/Group | Alisporivir
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug or Required Dose Reduction or Dose Interruption Due to Treatment-emergent Adverse Events
Time Frame: 48 weeks
Population: The study was terminated before the outcome measure time point.
Arm/Group | Alisporivir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (maximum exposure: 25 days) plus 30 days
Arm/Group | Alisporivir
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisporivir (N=6)
Nasopharyngitis (Infections and infestations) | 1
Pyrexia (General disorders) | 3
Headache (Nervous system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2
Chills (General disorders) | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Sleep Disorder (Psychiatric disorders) | 1
Asthenia (General disorders) | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study, none of the planned outcome measures could be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other